CLINICAL TRIAL: NCT03983161
Title: A Phase 1 Open-label, Single-dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Fedratinib in Subjects With Moderate and Severe Hepatic Impairment Compared With Healthy Subjects
Brief Title: A Pharmacokinetics and Tolerability Study of Fedratinib in Subjects With Moderate and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-CP-001; U1111-1233-7820 (Other: WHO)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers; Hepatic Impairment
Keywords: Healthy Subjects; Fedratinib; Hepatic impairment; Pharmacokinetics
MeSH Terms: interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fedratinib in moderate hepatic impairment subjects (Experimental): A single oral dose of 300 mg of fedratinib will be given to subjects with moderate hepatic impairment
  Interventions: Drug: Fedratinib
- Fedratinib in severe hepatic impairment subjects (Experimental): A single dose of 200 mg of fedratinib will be given to subjects with severe hepatic impairment
  Interventions: Drug: Fedratinib
- Fedratinib in healthy vs moderate hepatic impairment subjects (Experimental): A single oral dose of 300 mg of fedratinib will be given to healthy subjects with normal hepatic function.
  Interventions: Drug: Fedratinib
- Fedratinib in healthy vs severe hepatic impairment subjects (Experimental): A single oral dose of 200 mg of fedratinib will be given to healthy subjects with normal hepatic function.
  Interventions: Drug: Fedratinib

INTERVENTIONS:
Drug: Fedratinib — Fedratinib

SUMMARY:
This is a Phase 1, multicenter, nonrandomized, open-label, single oral dose study to assess the PK of fedratinib in subjects with moderate and severe hepatic impairment, and in matched subjects with normal hepatic function.

Degrees of hepatic impairment will be determined during screening by the subject's score according to Pugh's Modification of Child's Classification of Severity of Liver Disease.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all subjects (Groups 1 through 4)

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements, including the restrictions
3. Subject is male, or non-pregnant and non-nursing female ≥ 18 and ≤ 75 years of age at the time of signing the Informed Consent Form (ICF).
4. Subject has body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at screening.
5. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level in the post-menopausal range according to the laboratory used at Screening); FSH to be performed at the discretion of the Investigator in consultation with the Sponsor's Medical Monitor.
6. A female of childbearing potential (FCBP) must:

   1. Have a negative pregnancy test as verified by the Investigator at Screening and Baseline (prior to starting study treatment). She must agree to ongoing pregnancy testing during the course of the study, as applicable, and after the end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use, and be able to comply with, any one of the following highly effective contraception methods without interruption, beginning at least 14 days prior to dosing, during the study treatment, and for at least 30 days after the last dose of IP.

      * Hormonal contraception (eg, birth control pills, intravaginal ring, transdermal patch, injection, implant); intrauterine device (IUD); tubal ligation; or a partner with a vasectomy. The chosen form of birth control must be effective by the time the subject receives the first dose of IP.
7. Male subjects must:

   a. Practice true abstinence (which must be reviewed monthly, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made from natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while receiving study treatment, and for at least 30 days after the last dose of IP, even if he has undergone a successful vasectomy.
8. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator.
9. Subject is afebrile (febrile is defined as ≥ 38°C or 100.3°F), with supine systolic blood pressure (BP) ≥ 90 and ≤ 160 mm Hg, supine diastolic BP ≥ 50 and ≤ 100 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute at Screening.

   Inclusion Criteria for Subjects with Moderate or Severe Hepatic Impairment (Groups 1 and 3)

   Each subject with moderate or severe hepatic impairment must also meet all the criteria listed below for entry:
10. Subject has moderate or severe hepatic impairment or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
11. Subject has moderate (Group 1) or severe (Group 3) hepatic impairment as defined by Child-Pugh Score.

    * Group 1 subjects (moderate hepatic impairment) are required to have documented confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy, or imaging study with a Child-Pugh score of ≥ 7 to ≤ 9 at Screening.
    * Group 3 subjects (severe hepatic impairment) are required to have documented confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy, or imaging study with a Child-Pugh score of ≥ 10 to ≤ 13 at Screening.

    If biopsy or laparoscopy is not performed prior to Screening, subjects can be included only if they have chronic liver disease and objective evidence of portal hypertension (ascites diagnosis by imaging or varices), or current medication for consequences of portal hypertension.

    Subjects should be enrolled into the group corresponding to the Child-Pugh classification score that most accurately reflects the most severe hepatic disease classification within the past 6 months (based on past medical history or physical examination observation).

    *Note: If a Child-Pugh score was previously calculated and documented in the last 6 months, and it is more severe than the one calculated at Screening, then that previous value will be used for study entry purposes. If the Screening Child-Pugh score is more severe, then it will be used. If no score was calculated in the 6 months prior to Screening, then the score obtained at Screening will be used. Adequate documentation should be provided to substantiate the Child-Pugh score assigned to each subject.
12. Subject must be medically stable for at least 1 month before Screening with clinically acceptable medical history, PE, clinical laboratory tests, vital signs, and 12-lead ECGs consistent with the underlying stable hepatic impairment condition, as judged by the Investigator.
13. Subject must be stable on a concomitant medication regimen (defined as not starting a new medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 7 days or 5 half-lives [whichever is longer] before dosing with fedratinib).
14. Subject may be treated with diuretics for ascites. Subjects with severe ascites at time of enrollment may be included at the discretion of the Investigator.
15. Subject may have a history of encephalopathy; however, they must be on stable treatment for at least 1 month prior to Screening, and must not have had an acute encephalopathic episode in the 1 month prior to Screening.
16. Subjects must not have history of hepatorenal syndrome or hemolysis.
17. Subject has a normal or clinically acceptable 12-lead ECG at Screening (QTcF ≤ 480 msec).
18. Subject must have estimated creatinine clearance ≥ 60 mL/min at Screening as calculated by the Cockcroft-Gault formula.

    Inclusion Criteria for a Matched Healthy Subjects (Groups 2 and 4) Each matched healthy subject must meet all the criteria listed below for entry:
19. Subject is free of any clinically significant disease that would interfere with the study evaluations.
20. Subject has liver-related laboratory test results within the respective reference ranges or judged as clinically acceptable by the Investigator.
21. Subject must match a subject in Groups 1 or 3, as needed, with respect to sex, age (± 10 years), and weight (± 13.6 kg [30 pounds]).
22. Subject is in good health as determined by past medical history, PE, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (ie, hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the Investigator.
23. Subject has a normal or clinically acceptable 12-lead ECG at Screening. In addition:

    1. If male, subject has a QTcF value ≤ 450 msec at Screening.
    2. If female, subject has a QTcF value ≤ 470 msec at Screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has prior history of Wernicke's encephalopathy (WE).
2. Subject has signs or symptoms of WE (eg, severe ataxia, ocular paralysis or cerebellar signs) without documented exclusion of WE by thiamine level and brain MRI.
3. Subject has thiamine deficiency, defined as thiamine levels in whole blood below normal range according to institutional standard and not demonstrated to be corrected prior to enrollment into the study.
4. Subject has any significant and relevant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study at the Investigator's discretion.
5. Subject has any condition that places the subject at an unacceptable risk if he or she were to participate in the study.
6. Subject has any condition that confounds the ability to interpret data from the study.
7. Subject is pregnant or breastfeeding.
8. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever was longer).
9. Subject has used moderate or strong CYP3A4 and/or CYP2C19 inducers and/or inhibitors (including St. John's wort) within 14 days or 5 half-lives, whichever is longer, prior to the first dose administration. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP3A4 (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
10. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. Subjects with appendectomy and cholecystectomy may be included.
11. Subject donated blood or plasma within 2 weeks before dose administration to a blood bank or blood donation center.
12. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs.

    a. If positive drug screen in a subject with hepatic impairment is due to prescription drug use, the specific drug and dosing regimen of the prescription drug must be reviewed with the Sponsor's Medical Monitor to ensure lack of interference with the PK assessments of this study, according to the protocol. The decision and its rationale will be documented in the Trial Master File.
13. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 1 year before dose administration, or a positive alcohol screen.
14. Subject has had a positive result to the test for human immunodeficiency virus (HIV) antibodies at Screening.
15. Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
16. Subject has received live vaccination (excluding seasonal flu vaccination) within 90 days of dosing.
17. Subject is part of the clinical staff personnel or a family member of the study site staff.
18. Subject is, for any reason, deemed by the investigator to be inappropriate for this study, including a subject who is unable to communicate or to cooperate with the Investigator or the clinical staff.
19. Subject has a hypersensitivity to ondansetron. 4.3.1. Exclusion Criteria for Subjects with Moderate or Severe Hepatic Impairment (Groups 1 and 3) The presence of any of the following will exclude a hepatically-impaired subject from enrollment:
20. Subject has any serious medical condition (excluding hepatic impairment and related complications), clinically significant laboratory abnormality not related to hepatic impairment and related complications, or psychiatric illness that would prevent the subject from signing the ICF and participating in the study per Investigator discretion.
21. Subject has current hepatic encephalopathy with time- or place- disorientation, somnolence, stupor, coma, no personality/behavior, rigidity, or hyperactive reflexes - or has had such within 1 month of Screening. Hepatic subjects with history of grade 3 or 4 encephalopathy who are treated with concomitant medications to control encephalopathy will receive pre-treatment score for the Child-Pugh classification.
22. Subject has a history of incipient/planned liver transplantation within 6 months of Screening or has received a liver transplant.

    Exclusion Criteria for a Matched Healthy Subject (Groups 2 and 4) Each matched healthy subject will be excluded from entry if any of the criteria listed below are met:
23. Subject has any clinically significant laboratory abnormality that, in the opinion of the Investigator, is considered to prevent the subject from safely completing the study.
24. Subject has any unstable clinically significant illness within 3 months prior to the study.
25. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
26. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days or 5 drug half-lives (whichever is longer) prior to the first dose administration of fedratinib.

    a. A subject who has used (or will have used) a prescribed medication less than 30 days prior to (but at least 5 half-lives prior to) fedratinib dosing may be admitted into the study if such usage is not expected by the Investigator to have persistent PK effects at the time of fedratinib dosing. Such effects may include, but are not limited to, cytochrome induction or covalent cytochrome inhibition. These cases must be approved by Sponsor's Medical Monitor. The decision and its rationale will be documented in the Trial Master File.
27. Subject has used any nonprescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days or 5 drug half-lives (whichever is longer) prior to the first dose administration of fedratinib.

    a. A subject who has used (or will have used) a nonprescribed medication less than 14 days prior to (but at least 5 half-lives prior to) fedratinib dosing may be admitted into the study if such usage is not expected by the Investigator to have persistent PK effects at the time of fedratinib dosing. Such effects may include, but are not limited to, cytochrome induction or covalent cytochrome inhibition. These cases must be approved by Sponsor's Medical Monitor. The decision and its rationale will be documented in the Trial Master File.
28. Subject is known to have a history of hepatitis B and/or hepatitis C, or have a positive result to the test for HIV antibodies at screening Note: Subjects who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Fedratinib Pharmacokinetic (PK): AUC0-t | Up to approximately 8 days.
  Estimation of AUC from time zero to the last measured time point
Fedratinib Pharmacokinetic (PK): AUC0-∞ | Up to approximately 8 days.
  Estimation of AUC from time zero extrapolated to infinity
Fedratinib Pharmacokinetic (PK): Cmax | Up to approximately 8 days.
  Estimation of maximum observed plasma concentration
Fedratinib Pharmacokinetic (PK): Tmax | Up to approximately 8 days.
  Estimation of time to reach Cmax
Fedratinib Pharmacokinetic (PK): t1/2 | Up to approximately 8 days.
  Estimation of terminal elimination half-life
Fedratinib Pharmacokinetic (PK): CL/F | Up to approximately 8 days.
  Estimation of apparent total plasma clearance when dosed orally
Fedratinib Pharmacokinetic (PK): Vz/F | Up to approximately 8 days.
  Estimation of apparent volume of distribution when dosed orally

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 30 days after completion of study treatment
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm